CLINICAL TRIAL: NCT05814263
Title: Direct HIS/LBB Pacing as an Alternative to Biventricular Pacing in Patients With Symptomatic Heart Failure Despite Optimal Medical Treatment and ECG With Typical Left Bundle Branch Block
Brief Title: HIS Alternative II - UK Site
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22HH7978
Record Dates: First submitted 2023-03-16; First posted 2023-04-14 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Left Bundle-Branch Block
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the staff performing and evaluating echocardiography and hall-walk tests are blinded to the treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIS/LBB pacing (Experimental): In this arm a right ventricular (RV) lead or implantable cardioverter defibrillator (ICD) lead is placed first and then implantation of a HIS-pacing lead is attempted. If it is not possible to find and pace HIS, to correct the LBBB or the threshold for correcting the LBBB is > 2.5 V at 1 ms, implantation of a LBB-pacing lead is attempted instead. If that is not possible either, a left ventricular (LV) lead is implanted.
  Intervention: Device: HIS/LBB pacing
  Interventions: Device: HIS/LBB pacing
- LV pacing (Active Comparator): In this arm an RV-lead or ICD-lead is placed first and then implantation of a LV-pacing lead is attempted. If this is not possible due to anatomical difficulties (no coronary sinus (CS) access, no available branches other than v cordis anterior or v cordis media) or electrical difficulties (no capture below 4 V at 1.0 msec or phrenic nerve stimulation < 2x pacing threshold), implantation of a HIS-pacing lead is attempted instead. If that is not possible or the threshold for correcting the LBBB is > 2.5 V at 1 ms, implantation of a LBB-pacing lead is attempted instead.
  Intervention: Device: LV pacing
  Interventions: Device: LV pacing

INTERVENTIONS:
Device: HIS/LBB pacing — 3830 lead to HIS or LBB
  Arms: HIS/LBB pacing
Device: LV pacing — LV lead in a CS branch
  Arms: LV pacing

SUMMARY:
The study will investigate the feasibility of using direct HIS pacing or left bundle branch pacing (LBB pacing) as an alternative to biventricular pacing in patients with symptomatic heart failure and an ECG with a typical left bundle branch block pattern.

DETAILED DESCRIPTION:
Biventricular pacing has for more than a decade been standard of care for patients with HFrEF, LVEF < 35%, NYHA II-IV despite optimal medical treatment and an ECG with left bundle branch block (LBBB). However, it is not always ideal because of several drawbacks such as phrenic nerve capture, inability to reach late activated areas and many more. Direct HIS pacing can in many cases capture the left bundle and provide normal electrical activation of the left ventricle but sometimes with high pacing thresholds. Recently direct left bundle branch pacing has shown promise with synchronous activation of the left ventricle at low pacing thresholds.

In the present study the investigators randomize 125 patients in one center to either conventional CRT (45 patients) or HIS/LBB pacing (80 patients). In the HIS/LBB arm, direct HIS-pacing is attempted first but if its not possible or the pacing threshold for capturing the left bundle branch is > 2.5 V at 1 ms the investigators switch to placing a LBB-lead.

Power calculation for non-inferiority: With the 50 patients in the first His Alternative study (25 Biv-CRT og 25 His-CRT) the investigators observed a fall in systolic volumes of 34% and 46% with a standard deviation of 13-16%. Using these numbers it would take at least 108 patients to be 90% sure that the lower limit of a one-sided 97.5% confidence interval (equal to a 95% two-sided confidence interval) would be over the non-inferiority limit of -10%.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, ischemic or non-ischemic cardiomyopathy with LVEF ≤ 35% assessed by echocardiography, NYHA class II-IV heart failure symptoms despite optimal medical treatment and

  * Either planned new implantation of a biventricular pacing system (CRT-P or CRT-D), where the ECG is with sinus rhythm and a typical left bundle branch block (see definition below)
  * Or planned upgrade of an existing pacemaker or ICD to a biventricular pacing system (CRT-P or CRT-D), where the ECG is with sinus rhythm and a typical left bundle branch block or there has been> 90% right ventricular pacing from an existing pacemaker for at least 2 months prior to enrollment
* Signed informed consent
* Typical left bundle branch block:

  * QRS width > 130 msec for women and > 140 msec for men QS or rS pattern in leads V1 and V2, and mid-QRS plateau phase with or without extras in at least 2 of leads V1, V2, V5, V6, I, and aVL

Exclusion Criteria:

* Existing biventricular pacing system
* Permanent atrial fibrillation
* Severe renal failure with eGFR < 30 ml/min
* AMI or CABG within the last three months
* The patient does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Left ventricular end-systolic volume | 6 months
  Echocardiographic response after 6 months defined as decrease in left ventricular systolic volume of ≥ 15% of baseline
Success rate of implanting a HIS-bundle lead with capture of the left bundle branch or a LBB-lead with narrowing of QRS | 6 months
  The success rate of implanting a pacing lead to the HIS-bundle with capture of the left bundle at a threshold < 2.5 V at 1 ms or implantation of a LBB lead with narrowing of the QRS duration and maintaining this effect at 6 month follow-up

SECONDARY OUTCOMES:
Change in LVEF and left ventricular chamber dimensions | 6 months
  Echocardiographic response assessed by chamber dimensions and LVEF on a continuous scale
Change in 6-min hall-walk test | 6 months
  Functional response after 6 months defined as an increase in 6-min walking distance of ≥ 20% of the initial value
Change in NYHA class | 6 months
  Symptomatic response after 6 months defined as a fall in NYHA class of ≥ 1
Change in Minnesota Living with Heart Failure score | 6 months
  Change in well-being after 6 months defined as a decrease in Minnesota Living With Heart Failure score of ≥ 15% of baseline
Shortening of QRS duration | 6 months
  Shortening the duration of the QRS complex defined as the widest paced QRS complex rated at 12-lead ECG after 6 months
Change in NT-pro BNP value | 6 months
  Change in NT-pro BNP value
Complications | 6 months
  Device-related complications (periprocedural: electrode reoperation, pneumothorax, hemothorax, pericardial bleeding/tamponade and later (after 30 days post implantation): LV/HIS electrode reoperation, change of device due to battery depletion and infection requiring extraction).

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Will share data with international arm of the project NCT04409119
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 6 months following final recruitment